CLINICAL TRIAL: NCT04694885
Title: Quality of Life Improvement of Breast Cancer Patients During Chemotherapy With Structured Psychological Interventions
Brief Title: Quality of Life Improvement During Chemotherapy
Acronym: QoLMa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Schwegler (Other)
Responsible Party: Sponsor-Investigator, Christian Schwegler, Scientific Collaborator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QoLMa
Record Dates: First submitted 2020-12-18; First posted 2021-01-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Female; Chemotherapy Effect
Keywords: Breast cancer; Chemotherapy; Hypnotherapy; Hypnosis; Quality of life; Anxiety; Depression; Immunity; Dose-response effect
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: The study is a monocentric randomized controlled trial with two parallel arms. All participants will be recruited in the University Hospital Basel (CH). They must be adult, female, diagnosed with first time breast cancer and undergoing adjuvant or neo-adjuvant chemotherapy. During chemotherapy, the control group as well as the intervention group will be offered the standard of psycho-oncological care. This means they can chose how much psychological support they want to use. Additionally, participants in the intervention group participate in 10 structured sessions of hypnotherapy aimed to alleviate quality of life. These therapeutic sessions will take place approximately every two to three weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The control group will receive the standard of psycho-oncological care.
- Standard of Care + Structured Hypnotherapy (Experimental): The intervention group will receive the standard of psycho-oncological care plus 10 hypnotherapeutic sessions every two weeks.
  Interventions: Behavioral: Structured Hypnotherapy

INTERVENTIONS:
Behavioral: Structured Hypnotherapy — The Intervention includes 10 structured hypnotherapy sessions lasting 45 to 60 minutes. During hypnosis, patients reach a trance-like state comparable to a deep relaxation. The therapist guides the patient verbally and also communicates with the patient.
  Patients will be supported to use their own imagination without suggesting any imagery. By repeatedly asking what the patient is perceiving, and by verbally repeating what the patient is saying, the therapist can help the patient to go deeper into trance. In these trance states the patient learns to reduce negative side effects of the chemotherapy and increase the quality of life by activating both physical and mental resources using imagination and focusing on positive memories and feelings.
  Other Names: Structured Psychological Intervention; Hypnosis
  Arms: Standard of Care + Structured Hypnotherapy

SUMMARY:
This study is a randomized controlled trial, taking place at the University Hospital Basel (CH). It aims at the alleviation of breast cancer patients' life quality during chemotherapy.

The intervention group will participate in 10 sessions of structured hypnotherapy during the course of chemotherapy in addition to the standard of care. The control group will have access to the standard of care without any additional treatment. The main goal of the study is to investigate whether quality of life is higher among patients in the intervention group. Additionally, it will be analyzed if the interventions have a positive effect on chemotherapy side effects, symptoms of anxiety and depression and the immune system. Finally, the relative dose intensity (RDI) as well as treatment schedule adherence will be assessed.

There are no risks to be expected from the intervention itself. In the case of positive findings, the standard of psycho-oncological care can be updated by integrating structured hypnotherapeutic interventions into the treatment of patients with breast cancer.

DETAILED DESCRIPTION:
Background:

Breast cancer patients who undergo chemotherapy are likely to experience lower life quality, side effects like nausea and vomiting and symptoms of anxiety or depression. At the same time their immune system is down regulated by a stress reaction following cancer diagnosis and also by the chemotherapy itself. Decrease of several immune factors is associated with lower survival expectancy.

Hypnotherapy uses methods like relaxation, symptom-control techniques, imagination and working with inner resources. They can be used to bring positive change for patients both mentally as well as physically. Self-hypnosis techniques are used to bring back a feeling of self-efficacy which is impaired in most cancer patients who report to lose control over their body.

Emerging evidence shows the effectiveness of hypnotherapy in reducing side-effects of medical treatments and improve mental health and quality of life of cancer patients. It was shown that hypnotherapy has a positive effect on several immune factors. But up to now it is not clear if there is also a positive effect on the immune system during chemotherapy.

During Chemotherapy it is important that patients adhere as much as possible to the treatment schedule and to the optimal dosage. Due to chemotherapy side-effects or other reasons it happens regularly that treatment needs be delayed or dosage reduced which in turn lowers the efficiency of the chemotherapy.

Objectives:

This study is designed to evaluate if hypnotherapy has a positive effect on quality of life, side-effects of chemotherapy, symptoms of anxiety and depression, the immune system and the relative dose intensity (RDI) of female breast cancer patients during the course of chemotherapy.

Study Flow:

After patients have been diagnosed with primary breast cancer and were assigned to either adjuvant or neo-adjuvant chemotherapy they are asked if they want to participate in the study and are given all the necessary information and consent form. If they agree, they will be randomly assigned to either the control group or the intervention group following a computer generated randomization list. Before the first session of hypnotherapy they will be given the first questionnaires (T0). Those assigned to the intervention group will be contacted by a therapist to fix a date for the first session, if possible before the first chemotherapy cycle or shortly after the first cycle, when the side effects are not yet present. During 4,5 months, patients will receive 6 cycles of chemotherapy and 10 session of hypnotherapy. They will have access to the standard of psycho-oncological care during the study. The control group will not receive any Hypnotherapy but also has access to the standard of psycho-oncological care.

Measurement Points:

T0 (Baseline) = After diagnosis and before the first chemotherapy cycle

T1 = First cycle of chemotherapy

T2 = Second cycle

T3 = Third cycle

T4 = Fourth cycle

T5 = Fifth cycle

T6 = Sixth cycle

The duration of one cycle will be approx. 3 weeks, depending on the individual chemotherapy regimen.This means that the total time for the chemotherapy of one patient will last around 18 weeks.

There are no risks to be expected from the intervention itself. In the case of positive findings, the standard of psycho-oncological care can be updated by integrating structured hypnotherapeutic interventions into the treatment of patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age 18 years
* Female
* Primary breast cancer
* Receiving neo-adjuvant or adjuvant chemotherapy

Exclusion Criteria:

* Verbal or cognitive deficits that are not compatible with outpatient psychotherapy
* Not consenting patients and vulnerable persons
* Psychological disorders that prevent patients from participating in the study (e.g. psychotic disorder)
* acute suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Average Summary Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 6 times within 18 weeks + baseline at day 1
  The outcome measure will be the average of all 6 time points on the EORTC QLQ-C30 summary score. The summary score ranges from 0 to 100 with higher scores representing a better quality of life. In the statistical analysis this average summary score will be corrected for values of the summary score at T0.

SECONDARY OUTCOMES:
Summary Score of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 7 times within 18 weeks
  Summary score of the EORTC QLQ-C30 on all 7 time points including baseline. The summary score ranges from 0 to 100 with higher scores representing a better quality of life. In the statistical analysis the summary score will be compared between all time points to see the development of life quality throughout the chemotherapy.
Side Effects of Chemotherapy | 7 times within 18 weeks
  Side effects of chemotherapy will also be captured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). It contains three symptom scales (fatigue, pain, nausea and vomiting) and single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation, diarrhea and financial problems). All symptom scales range from 1-4 with higher values representing higher levels of symptoms.
Hamilton Anxiety and Depression Scale - German Version (HADS-D) | 7 times within 18 weeks
  The HADS-D has two sub-scales for anxiety and depression. Each sub-scale ranges from 0 to 21 with higher values representing more severe symptoms of depression and anxiety respectively.
  <= 7 unproblematic
  8 - 10 threshold
  >= 11 problematic
Immune Factors | 3 times within 18 weeks
  Count of cells per micro-liter (μL) of:
  1. Natural killer cells (NK)
  2. CD4 (also called T-helper cells)
  3. CD8 (marker for cytotoxic T-cells)
Interleukin-6 | 3 times within 18 weeks
  Counts of picogram per milliliter (pg/mL) of IL-6 (interleukin-6)
Tumor Marker CA 15-3 | 3 times within 18 weeks
  Counts of international units per milliliter (IU/mL) of tumor marker CA 15-3
Relative Dose Intensity (RDI) | 18 weeks
  RDI = % dose x (planned days / used days). Reference values: >85% effective treatment, <=85% ineffective and significantly decreased survival chances.
Schedule Modification: Delayed Cycles | 18 weeks
  Delayed cycles. Reference value >=2. The less cycles are delayed, the more efficient is the chemotherapy. If two or more cycles have been delayed, we consider it a significant decrease in schedule adherence.
Schedule modification: Delayed Days | 18 weeks
  Delayed days. Reference value >=14. The less days are delayed, the more efficient is the chemotherapy. If 14 or more days have been delayed, we consider it a significant decrease in schedule adherence.

OTHER OUTCOMES:
Exploratory Analysis of the Correlation between Quality of Life, Anxiety, Depression and Immunfaktors and Tumor Marker | 18 weeks
  Individual correlations between quality of life, side effects of chemotherapy, anxiety and depression (specified as outcome measures 2 - 4) and each of the immune factors and tumor marker (outcome measures 5 - 7). Due to lack of pre-existing evidence, we make no predictions about direction and magnitude of the effects.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Ge, Dr., Study Director — University Hospital, Basel, Switzerland; Christian Schwegler, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual request will be evaluated and shared if appropriate.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of first results. Data will be available for 10 years.
Access Criteria: Will be evaluated upon request.